CLINICAL TRIAL: NCT06817590
Title: Nucleoside Therapy in Patients With Telomere Biology Disorders
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suneet Agarwal (Other)
Responsible Party: Sponsor-Investigator, Suneet Agarwal, Physician, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00049530
Record Dates: First submitted 2025-01-30; First posted 2025-02-10 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Telomere Biology Disorders; Dyskeratosis Congenita; Revesz Syndrome; Hoyeraal Hreidarsson Syndrome; Telomere Biology Disorders With Bone Marrow Failure; Interstitial Lung Disease Due to Systemic Disease (Telomere Biology Disorder); Pulmonary Fibrosis, Familial (Telomere Biology Disorder)
Keywords: nucleoside; phase I; deoxycytidine; deoxythymidine; telomere biology disorders; safety; tolerability; pharmacokinetics; telomere lengths; bone marrow; clonal hematopoiesis; bone marrow failure; pulmonary fibrosis
MeSH Terms: conditions — Dyskeratosis Congenita; Revesz Debuse syndrome; Hoyeraal Hreidarsson syndrome; Pulmonary Fibrosis; Bone Marrow Failure Disorders | interventions — Deoxycytidine; Thymidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- dC/dT (Experimental): Participants will take study therapy three times daily over 24 weeks with dose escalation.
  Interventions: Drug: deoxycytidine; Drug: deoxythymidine

INTERVENTIONS:
Drug: deoxycytidine — Oral administration, in combination with deoxythymidine
  Other Names: dC
Drug: deoxythymidine — Oral administration, in combination with deoxycytidine
  Other Names: thymidine; dT

SUMMARY:
The goal of this clinical trial is to learn if a combination therapy of deoxycytidine (dC) plus deoxythymidine (dT) is safe in patients with telomere biology disorders. The main questions it aims to answer are:

* Is the therapy safe with tolerable side effects in patients with telomere biology disorders?
* Are problems with the bone marrow or blood or lungs changed after 6 months of dC+dT treatment in patients with telomere biology disorders?

Participants will:

* Take study drug by mouth three times daily for 24 weeks
* Make approximately 2 visits to Boston Children's Hospital during the 24 weeks: once at the beginning of treatment and once at the end of treatment.
* Go to a lab for a blood draw an additional 6 times during treatment.
* Have 9 phone calls with a research nurse, including one 4 weeks after treatment ends.
* Keep a diary to track doses of study drug that were taken or missed.

DETAILED DESCRIPTION:
This is an investigator-initiated, single-arm, single-center phase 1 clinical trial investigating nucleoside therapy in patients telomere biology disorder (TBDs). TBDs are a group of rare, inherited conditions characterized by critically short telomeres which can limit cellular replication resulting in a wide spectrum of clinical manifestations. From a hematologic standpoint, patients with TBDs often present with bone marrow failure. Therapy options for bone marrow failure for patients with TBDs are limited to androgen therapy and hematopoietic cell transplantation, which are associated with significant challenges and toxicities. From a pulmonary standpoint, patients with TBDs can present with low oxygen levels due to hepatopulmonary syndrome or lung fibrosis, which requires organ transplantation. New therapeutic approaches are needed in patients with an underlying TBD. Recent studies emerging from multiple independent human genetic studies have established a critical role for deoxythymidine (dT) metabolism in human telomere maintenance and demonstrated that upregulation of nucleotide metabolism by dT supplementation in vitro led to telomere elongation. The goals of this trial are to (1) assess the safety and tolerability of enteral nucleoside therapy in patients with TBDs and (2) explore the clinical and biologic effects of enteral nucleoside therapy in patients with TBDs. A total of 36 pediatric and adult patients with a diagnosis of a TBD will be enrolled at Boston Children's Hospital. Patients will receive enteral nucleoside therapy for a total of 24 weeks. Drug diary reviews and safety and tolerability assessments will be conducted on a weekly basis during an initial dose-escalation phase (4 weeks) and then monthly until study treatment completion at week 24. Pharmacokinetic studies will be conducted on a subset of participants. Additionally, changes in lymphocyte telomere lengths, peripheral blood counts, bone marrow cellularity, clonal hematopoiesis, pulmonary function tests, and chest CT imaging may be explored pre- and post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 1 year and ≤ 70 years
* Karnofsky performance status ≥ 50 for participants ≥16 years of age and Lansky performance status ≥ 50 for participants <16 years of age
* Diagnosis requirement. Participants must meet at least one of the following requirements for a diagnosis of a telomere biology disorder:

  1. Age-adjusted mean telomere length < 1%ile in peripheral blood lymphocytes by flow cytometry-fluorescence in situ hybridization (flow-FISH), as reported by a Clinical Laboratory Improvement Amendments (CLIA)-approved laboratory

     OR
  2. Pathogenic or likely pathogenic variant(s) in one of the follow telomere biology associated genes: DKC1, TERC, TERT, NOP10, NHP2, WRAP53/TCAB1, TINF2, CTC1, RTEL1, ACD, PARN, NAF1, STN1, ZCCHC8, POT1, RPA1, DCLRE1B, TYMS, as reported by a CLIA-approved laboratory.
* Participants must exhibit at least one active clinical manifestation associated with a telomere biology disorder, in the judgment of the PI, which includes but is not limited to the following: one or more peripheral blood cytopenias, bone marrow hypocellular for age, pulmonary abnormalities, liver abnormalities, gastrointestinal bleeding, immunodeficiency or immune dysregulation, ophthalmologic abnormalities, or neurologic abnormalities.
* Participants must be able to take enteral liquids by mouth or enteral feeding tube.
* Female participants who are sexually active and could become pregnant must use two effective methods of contraception, at least one of which must be considered a highly effective method.
* Participants (or parent/legally authorized representative for minors) must demonstrate the ability to understand and willingness to provide informed consent, which will be documented using an institutionally approved informed consent procedure.

Exclusion Criteria:

* Participants must not have very severe aplastic anemia necessitating bone marrow transplant at the time of enrollment. Very severe aplastic anemia is defined by the presence of at least 2 of the following: ANC <200 cells/microliter, platelets <20,000 cells/microliter, absolute reticulocyte count <40,000 cells/microliter. If individuals with very severe aplastic anemia are not expected to undergo bone marrow transplant either due to the lack of an acceptable donor or medical co-morbidities and otherwise meet the inclusion/exclusion criteria, then they would be eligible for enrollment in this trial.
* Participants must not otherwise be expected to undergo bone marrow transplantation within 6 months of enrollment.
* Participants must not be taking concurrent medications intended to improve hematopoiesis such as androgens or growth factors, including granulocyte colony stimulating factor, erythropoietin, or thrombopoietin mimetics. If any of these therapies were taken previously, patients must wait 30 days after cessation of the therapy before enrollment on this trial.
* Participants must not have chronic diarrhea or an average baseline stool output of more than 4 stools per day.
* Participants must not have gastrointestinal disorders that may impair enteral absorption of dC/dT, such as inflammatory bowel disease or short bowel syndrome.
* Participants must not have chronic kidney disease with an estimated glomerular filtration rate < 60 mL/min/1.73 m2.
* Participants must not be on other medications or study agents or have other uncontrolled intercurrent illness that could interfere with study interpretation, in the opinion of the study Principal Investigator (PI)
* Participants must not have high-risk myelodysplastic syndrome or leukemia or other active malignancy.
* Pregnant individuals will not be eligible for enrollment given the physiological changes in blood counts that occur during pregnancy.
* Breastfeeding mothers will not be eligible for enrollment due to the unknown risk to nursing infants.

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related diarrhea [Tolerability] | 8 weeks from study drug initiation
  Proportion of study participants with grade 3 or higher treatment-related diarrhea refractory to dose adjustments
Incidence of treatment-related adverse events [Safety] | 8 weeks from study drug initiation
  Proportion of patients with grade 3 or higher treatment-related adverse events refractory to dose adjustments

SECONDARY OUTCOMES:
Change in hemoglobin | From pre-treatment baseline to end of treatment
  Change in hemoglobin (in grams per deciliter)
Change in platelet count | From pre-treatment baseline to end of treatment
  Change in platelet count (in thousands of cells per microliter)
Change in absolute neutrophil count | From pre-treatment baseline to end of treatment
  Change in absolute neutrophil count (in thousands of cells per microliter)
Maximal plasma concentration [Cmax] of dC | 24 weeks
  Maximal plasma concentration [Cmax] of dC will be obtained during pharmacokinetic profiling of dC at starting dose and maximum dose in some subjects
Maximal plasma concentration [Cmax] of dT | 24 weeks
  Maximal plasma concentration [Cmax] of dT will be obtained during pharmacokinetic profiling of dT at starting dose and maximum dose in some subjects
Plasma half-life [T1/2] of dC | 24 weeks
  Plasma half-life [T1/2] of dC will be obtained during pharmacokinetic profiling of dC at starting dose and maximum dose in some subjects
Plasma half-life [T1/2] of dT | 24 weeks
  Plasma half-life [T1/2] of dT will be obtained during pharmacokinetic profiling of dC at starting dose and maximum dose in some subjects

OTHER OUTCOMES:
Change in forced vital capacity (FVC) | Up to 24 weeks
  Change in forced vital capacity (percent predicted) on pulmonary function testing
Change in diffusing capacity of the lungs for carbon monoxide (DLCO) | Up to 24 weeks
  Change in diffusing capacity of the lungs for carbon monoxide (percent predicted) by pulmonary function testing

CONTACTS AND LOCATIONS:
Overall Officials: Helen Reed, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Childrens Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mannherz W, Agarwal S. Thymidine nucleotide metabolism controls human telomere length. Nat Genet. 2023 Apr;55(4):568-580. doi: 10.1038/s41588-023-01339-5. Epub 2023 Mar 23. PMID 36959362